CLINICAL TRIAL: NCT04876690
Title: Quality of Life of Crohn's Disease Patients With Complex Perianal Fistulas: an Observational, Cross-sectional Study
Brief Title: A Study of the Quality of Life in Adults With Crohn's Disease With Complex Perianal Fistulas
Acronym: CONFLICT
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: IBD-5007
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-02

CONDITIONS: Crohn Disease; Rectal Fistula
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease; Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CD Participants With CPF: Participants diagnosed with CD and CPF in the Portuguese routine clinical practice were assessed. Retrospective data on healthcare resource utilization related with CPF management in the previous three years was obtained from the medical records.

SUMMARY:
The main aim of the study is to assess the quality of life of people with Crohn's disease after treatment for complex perianal fistulas (CPF) in a standard clinic setting.

Study doctors will review the participants' medical records in the last 3 years. Participants will also be asked to visit the clinic once to complete 1 questionnaire on their quality of life.

DETAILED DESCRIPTION:
This is a national, observational, cross-sectional study. The study will assess the general QoL among CD participants with CPFs in the Portuguese routine clinical practice.

This study will enroll approximately 80 participants. All participants will be enrolled in one observational cohort.

The data will be collected retrospectively, from the medical records, on healthcare resource utilization and on the pharmacological and surgical treatments used for the management of CPFs in the three years prior to the inclusion visit.

This multi-center trial will be conducted in Portugal. The overall duration of this study is approximately 8 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with CD.
2. Presence of CPF(s), defined as >=1 of the following criteria:

   * High intersphincteric, high transsphincteric, extrasphincteric, or suprasphincteric location;
   * >=2 external openings;
   * Associated collections.
3. Attending routine gastroenterology appointments at the participating hospitals.

Exclusion Criteria:

1. Diagnosed with ulcerative colitis or indeterminate inflammatory bowel disease (IBD).
2. With non-complex fistulas or with fistulas types other than perianal (example, rectovaginal).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with CD and CPFs in the Portuguese routine clinical practice will be assessed.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- Portugal (5):
  - Centro Hospitalar e Universitario de Coimbra (CHUC), Coimbra
  - Centro Hospitalar Universitario de Lisboa Central (CHULC), Lisbon
  - Centro Hospitalar Universitario Lisboa Norte - Hospital de Santa Maria (CHULN-HSM), Lisbon
  - Centro Hospitalar Universitario de Sao Joao (CHUSJ), Porto
  - Centro Hospitalar Tondela-Viseu (CHTV), Viseu

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/6094ffc1ef0b71001e743c53

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data from participants were collected for this cross-sectional, observational study with a retrospective component at two investigative sites in Portugal from 9 July 2021 to 27 May 2022.
Pre-assignment Details: Participants with a diagnosis of Crohn's disease (CD) with complex perianal fistulas (CPF) were enrolled from the investigative sites' database and were observed in a cross-sectional way along with a retrospective component to collect data for healthcare resource utilization and on the pharmacological and surgical treatments in this study.
Period: Overall Study
Arm/Group | CD Participants With CPF
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CD Participants With CPF
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.40 (12.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Portugal | 15
Height [Mean (Standard Deviation); unit: centimeter] | 168.60 (8.28)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 68.45 (12.05)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/meter^2] — BMI=Weight (kg)/Height (meter)^2
  kg/meter^2 | 24.11 (4.11)

OUTCOME MEASURES:

1. Primary Outcome: Meta-Scores of the 12-Item Short Form Health Survey (SF-12) Questionnaire's Physical Component Score [PCS-12]
Description: SF-12 is 12-item self-report that assesses physical and mental health related general quality of life (QoL) whose results are expressed in terms of two meta-scores: the physical component summary (PCS) and the mental component summary (MCS), of which the PCS component is presented in this outcome measure. The PCS score has a range of 0 to 100. Higher scores indicate better physical functioning.
Time Frame: At inclusion visit (Day 1)
Population: All eligible participants with CD and CPAF were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CD Participants With CPF
Number analyzed (Participants) | 15
score on a scale | 45.36 (7.58)

2. Primary Outcome: Meta-Scores of the SF-12 Questionnaire's Mental Component Score [MCS-12])
Description: SF-12 is 12-item self-report that assesses physical and mental health related general quality of life (QoL) whose results are expressed in terms of two meta-scores: the PCS and the MCS, of which the MCS component is presented in this outcome measure. The MCS score has a range of 0 to 100. Higher scores indicate better mental functioning.
Time Frame: At inclusion visit (Day 1)
Population: All eligible participants with CD and CPAF were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CD Participants With CPF
Number analyzed (Participants) | 15
score on a scale | 38.00 (8.48)

3. Secondary Outcome: Short Inflammatory Bowel Disease Questionnaire (SIBDQ) Score
Description: The SIBDQ is an instrument used to assess QoL and is a disease-specific health-related quality of life questionnaire, that consists of 10 questions, each question is scored on a scale from 1 (poor quality of life) to 7 (good quality of life). The total score is reported and ranges from 10 to 70 with a higher score indicating a better health-related QoL.
Time Frame: At inclusion visit (Day 1)
Population: All eligible participants with CD and CPAF were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CD Participants With CPF
Number analyzed (Participants) | 15
score on a scale | 45.00 (10.72)

4. Secondary Outcome: Sexual Quality of Life-Male (SQOL-M) Questionnaire Score for Male Participants
Description: SQOL-M assessed the relationship between male sexual dysfunction and quality of life. It contains 11 items, each items are scored from 1 to 6 points (worst to best), completely agree = 1 to completely disagree = 6. The total score can range from 11 to 66 points. Higher scores indicate better male sexual quality of life.
Time Frame: At inclusion visit (Day 1)
Population: All eligible male participants with CD and CPAF were included in the analysis and are presented as the overall number of participants analyzed in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CD Participants With CPF
Number analyzed (Participants) | 7
score on a scale | 44.57 (14.59)

5. Secondary Outcome: Sexual Quality of Life-Female (SQOL-F) Questionnaire Score for Female Participants
Description: SQOL-F assessed the relationship between female sexual dysfunction and quality of life. It consists of 18 items, rated using a six-point scale (completely agree to completely disagree). The total score can range from 18 to 108 points. Higher scores indicate better female sexual quality of life.
Time Frame: At inclusion visit (Day 1)
Population: All eligible female participants with CD and CPAF with data available for analyses were included and are presented as the overall number of participants analyzed in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CD Participants With CPF
Number analyzed (Participants) | 5
score on a scale | 72.80 (25.54)

6. Secondary Outcome: Fecal Incontinence as Assessed by Wexner Score
Description: Fecal incontinence is measured by Wexner score. It consists of five questions to assess the degree of incontinence (solid, liquid, gas, wears pad, lifestyle alteration). The frequency of each type of incontinence is rated on a scale ranging from 0 (never) to 4 (always or to once a day) so that the sum of the frequencies add up to a total score that ranges from 0 to 20. Higher scores indicate worse fecal incontinence.
Time Frame: At inclusion visit (Day 1)
Population: All eligible participants with CD and CPAF were included in the analysis. Overall number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CD Participants With CPF
Number analyzed (Participants) | 14
score on a scale | 7.43 (5.50)

7. Secondary Outcome: Work Productivity and Activity Impairment (WPAI) as Assessed by WPAI Questionnaire Score
Description: WPAI score was used to describe the indirect healthcare resources. It is self-administered 6-item questionnaire (scale of 0-10) which assesses the effect of disease on work productivity in the past 7 days obtained for absenteeism (work time missed), presenteeism (impairment at work / reduced on-the-job effectiveness), work productivity loss (overall work impairment / absenteeism plus presenteeism) and activity impairment / disability. Scores are presented as percentages (multiplying the scores by 100), Domain scores are expressed as a percentage, with a range of scores form 0-100%, with 0% representing no impact on productivity and 100% representing complete impact on productivity. Higher scores indicate greater impairment.
Time Frame: At inclusion visit (Day 1)
Population: All eligible participants with CD and CPAF were included in the analysis. Number analyzed is the number of participants with data available for analysis in the specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CD Participants With CPF
Number analyzed (Participants) | 15
score on a scale
  Absenteeism: number analyzed (Participants) | 9
  Absenteeism | 3.80 (6.85)
  Presenteeism: number analyzed (Participants) | 9
  Presenteeism | 57.78 (29.91)
  Work Productivity Loss: number analyzed (Participants) | 9
  Work Productivity Loss | 58.89 (30.28)
  Activity Impairment | 52.67 (31.27)

8. Secondary Outcome: Number of Participants Characterized Based on Healthcare Resource Utilization (HCRU) Within Previous 3 Years
Description: Number of participants characterized based on HCRU associated with complex perianal fistulas (CPFs) management within the three years prior to the inclusion visit were collected. HCRU includes gastroenterology and other medical specialty appointments for the management of CPF; emergency room visits due to CPF; hospitalizations (greater than or equal to [>=] 24 hours) due to CPF, and intensive care unit (ICU) admission. Only categories with at least one participant with event are reported.
Time Frame: Up to 3 years prior to the inclusion visit at Day 1
Population: All eligible participants with CD and CPAF were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CD Participants With CPF
Number analyzed (Participants) | 15
Participants
  Any Medical Specialty Appointments for the Management of CPF | 15
  Emergency Room Visits due to CPF | 3
  Hospitalizations (>= 24 Hours) due to CPF | 5

9. Secondary Outcome: Number of Participants Categorized Based on Sociodemographic and Anthropometric Characteristics
Description: Sociodemographic and anthropometric variables included age (in years), sex (male or female), and body mass index (BMI).
Time Frame: At inclusion visit (Day 1)
Population: All eligible participants with CD and CPAF were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CD Participants With CPF
Number analyzed (Participants) | 15
Participants
  Age: 22 to 64 Years | 15
  Sex: Female | 8
  Sex: Male | 7
  BMI: Underweight | 0
  BMI: Normal range | 9
  BMI: Overweight | 4
  BMI: Obese | 2

10. Secondary Outcome: Number of Participants With Moderate to Severe Crohn's Disease (CD) Stratified by Clinical Characteristics
Description: The Montreal classification index for CD is used to classify the extent of the disease activity. It consists of two parameters: location and behavior of the disease activity. There are four different disease locations presented: Location 1 (L1) is ileum, Location 2 (L2) is colonic disease, Location 3 (L3) is ileocolon and Location 4 (L4) is isolated upper gastrointestinal (GI) tract disease. The first three categories (L1-L3) is combined with L4 where disease sites coexisted. There are 4 different categories for the behavior of the disease activity: Behavior 1 (B1) is non stenosing or non penetrating; Behavior 2 (B2) was stenosing; Behavior 3 (B3) is penetrating and p as perianal disease (p). The first 3 categories (B1 to B3) could be added with p to indicate coexisting perianal disease. Perianal disease (p) is defined as the presence of perianal abscesses or fistulae.
Time Frame: At inclusion visit (Day 1)
Population: All eligible participants with CD and CPAF were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CD Participants With CPF
Number analyzed (Participants) | 15
Participants
  Disease Location 1: Terminal Ileum | 4
  Disease Location 1 + 4: Terminal Ileum + Upper Gastrointestinal | 1
  Disease Location 2: Colon | 3
  Disease Location 3: Ileocolon | 5
  Disease Location 3 + 4: Ileocolon + Upper Gastrointestinal | 2
  Disease Behavior, Perianal Disease B1p: Nonstricturing, Nonpenetrating + Perianal | 8
  Disease Behavior, Perianal Disease B2p: Stricturing + Perianal | 5
  Disease Behavior, Perianal Disease B3p: Penetrating + Perianal | 2

11. Secondary Outcome: Number of Participants Characterized Based on Pharmacological Treatments and Surgeries for CPF
Description: For each pharmacological treatment (antibiotics, monoclonal antibodies, immunosuppressants, and others), participants were divided into three categories (current users, past users, and non-users) considering the three years prior to the inclusion visit. Surgical treatment in the last three years for the management of CPF was also recorded. A participant may be included in more than one category.
Time Frame: Up to 3 years prior to the inclusion visit at Day 1
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | CD Participants With CPF
Number analyzed (Participants) | 15
Participants
  Current Users: Antibiotics: number analyzed (Participants) | 14
  Current Users: Antibiotics | 2
  Current Users: Monoclonal Antibodies: number analyzed (Participants) | 14
  Current Users: Monoclonal Antibodies | 13
  Current Users: Immunosuppressants: number analyzed (Participants) | 14
  Current Users: Immunosuppressants | 7
  Past Users: Antibiotics: number analyzed (Participants) | 11
  Past Users: Antibiotics | 10
  Past Users: Monoclonal Antibodies: number analyzed (Participants) | 11
  Past Users: Monoclonal Antibodies | 2
  Past Users: Immunosuppressants: number analyzed (Participants) | 11
  Past Users: Immunosuppressants | 2
  Non-users: Antibiotics | 5
  Non-users: Monoclonal Antibodies | 2
  Non-users: Immunosuppressants | 7
  Non-users: Others | 15
  Surgical Treatment in the Last Three Years for the Management of CPF- Yes: number analyzed (Participants) | 12
  Surgical Treatment in the Last Three Years for the Management of CPF- Yes | 11
  Surgical Treatment in the Last Three Years for the Management of CPF- No: number analyzed (Participants) | 12
  Surgical Treatment in the Last Three Years for the Management of CPF- No | 1

12. Secondary Outcome: Correlation Between General QoL PCS-12 and the Participants Socio-demographic, Anthropometric and Clinical Characteristics Assessed as PCS Score Stratified Based on Qualitative Variables
Description: The following qualitative variables were considered for the bivariate analysis: sex, smoking status, employment status, extraintestinal manifestations of Crohn's disease, Montreal classification for CD disease (age at onset, disease location, and disease behavior), fistula type and position, CD disease activity, treatment-naïve, surgery-naïve, type of surgery, and presence of seton, perianal abscess and anorectal stricture. PCS-12 scores were transformed to a 0 to 100, with higher scores indicating better quality of life.
Time Frame: At inclusion visit (Day 1)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CD Participants With CPF
Number analyzed (Participants) | 15
score on a scale
  PCS-12: Sex- Male: number analyzed (Participants) | 7
  PCS-12: Sex- Male | 48.63 (8.16)
  PCS-12: Sex- Female: number analyzed (Participants) | 8
  PCS-12: Sex- Female | 42.50 (6.15)
  PCS-12: Employment Status- Employed: number analyzed (Participants) | 9
  PCS-12: Employment Status- Employed | 44.01 (7.33)
  PCS-12: Employment Status- Unemployed: number analyzed (Participants) | 3
  PCS-12: Employment Status- Unemployed | 48.22 (12.30)
  PCS-12: Employment Status- Retired: number analyzed (Participants) | 2
  PCS-12: Employment Status- Retired | 48.18 (3.49)
  PCS-12: Employment Status- Student: number analyzed (Participants) | 1
  PCS-12: Employment Status- Student | 43.25 (NA) — Standard deviation (SD) was not estimable due to low number of participants with event.
  PCS-12: Employment Status- Other: number analyzed (Participants) | 0
  PCS-12: Smoking Status- Never: number analyzed (Participants) | 8
  PCS-12: Smoking Status- Never | 47.90 (7.66)
  PCS-12: Smoking Status- Former: number analyzed (Participants) | 2
  PCS-12: Smoking Status- Former | 45.08 (0.42)
  PCS-12: Smoking Status- Current: number analyzed (Participants) | 5
  PCS-12: Smoking Status- Current | 41.40 (8.12)
  PCS-12: Age at Onset of CD Diagnosis - At or Below 16 Years: number analyzed (Participants) | 1
  PCS-12: Age at Onset of CD Diagnosis - At or Below 16 Years | 45.37 (NA) — Standard deviation (SD) was not estimable due to low number of participants with event.
  PCS-12: Age at Onset of CD Diagnosis - Between 17 and 40 Years: number analyzed (Participants) | 10
  PCS-12: Age at Onset of CD Diagnosis - Between 17 and 40 Years | 45.22 (9.06)
  PCS-12: Age at Onset of CD Diagnosis - Above 40 Years: number analyzed (Participants) | 4
  PCS-12: Age at Onset of CD Diagnosis - Above 40 Years | 45.70 (4.70)
  PCS-12: Disease Location 1- Terminal Ileum: number analyzed (Participants) | 4
  PCS-12: Disease Location 1- Terminal Ileum | 54.14 (4.46)
  PCS-12: Disease Location 1 + 4- Terminal Ileum + Upper Gastrointestinal: number analyzed (Participants) | 1
  PCS-12: Disease Location 1 + 4- Terminal Ileum + Upper Gastrointestinal | 43.25 (NA) — Standard deviation (SD) was not estimable due to low number of participants with event.
  PCS-12: Disease Location 2- Colon: number analyzed (Participants) | 3
  PCS-12: Disease Location 2- Colon | 41.14 (4.28)
  PCS-12: Disease Location 2 + 4- Colon + Upper Gastrointestinal: number analyzed (Participants) | 0
  PCS-12: Disease Location 3- Ileocolon: number analyzed (Participants) | 5
  PCS-12: Disease Location 3- Ileocolon | 43.64 (6.87)
  PCS-12: Disease Location 3 + 4- Ileocolon + Upper Gastrointestinal: number analyzed (Participants) | 2
  PCS-12: Disease Location 3 + 4- Ileocolon + Upper Gastrointestinal | 39.47 (8.34)
  PCS-12: Disease Location 4- Upper Gastrointestinal: number analyzed (Participants) | 0
  PCS-12: Disease Behavior- Nonstricturing, Nonpenetrating + Perianal: number analyzed (Participants) | 8
  PCS-12: Disease Behavior- Nonstricturing, Nonpenetrating + Perianal | 44.25 (7.33)
  PCS-12: Disease Behavior- Stricturing + Perianal: number analyzed (Participants) | 5
  PCS-12: Disease Behavior- Stricturing + Perianal | 47.61 (9.16)
  PCS-12: Disease Behavior- Penetrating + Perianal: number analyzed (Participants) | 2
  PCS-12: Disease Behavior- Penetrating + Perianal | 44.15 (7.40)
  PCS-12: Extraintestinal Manifestation of CD- Yes: number analyzed (Participants) | 2
  PCS-12: Extraintestinal Manifestation of CD- Yes | 49.37 (12.60)
  PCS-12: Extraintestinal Manifestation of CD- No: number analyzed (Participants) | 13
  PCS-12: Extraintestinal Manifestation of CD- No | 44.74 (7.13)
  PCS-12: Fistula With High Intersphincteric Type- Yes: number analyzed (Participants) | 3
  PCS-12: Fistula With High Intersphincteric Type- Yes | 50.72 (7.52)
  PCS-12: Fistula With High Intersphincteric Type- No: number analyzed (Participants) | 12
  PCS-12: Fistula With High Intersphincteric Type- No | 44.02 (7.29)
  PCS-12: Fistula With High Transsphincteric Type- Yes: number analyzed (Participants) | 3
  PCS-12: Fistula With High Transsphincteric Type- Yes | 41.58 (3.37)
  PCS-12: Fistula With High Transsphincteric Type- No: number analyzed (Participants) | 12
  PCS-12: Fistula With High Transsphincteric Type- No | 46.30 (8.14)
  PCS-12: Fistula With Suprasphincteric Type- Yes: number analyzed (Participants) | 2
  PCS-12: Fistula With Suprasphincteric Type- Yes | 38.08 (1.18)
  PCS-12: Fistula With Suprasphincteric Type- No: number analyzed (Participants) | 13
  PCS-12: Fistula With Suprasphincteric Type- No | 46.48 (7.54)
  PCS-12: Fistula With Extrasphincteric Type- Yes: number analyzed (Participants) | 2
  PCS-12: Fistula With Extrasphincteric Type- Yes | 39.64 (8.58)
  PCS-12: Fistula With Extrasphincteric Type- No: number analyzed (Participants) | 13
  PCS-12: Fistula With Extrasphincteric Type- No | 46.24 (7.39)
  PCS-12: Fistula With Superficial Type- Yes: number analyzed (Participants) | 0
  PCS-12: Fistula With Superficial Type- No | 45.36 (7.58)
  PCS-12: Fistula With Low Intersphincteric Type- Yes: number analyzed (Participants) | 2
  PCS-12: Fistula With Low Intersphincteric Type- Yes | 54.65 (3.94)
  PCS-12: Fistula With Low Intersphincteric Type- No: number analyzed (Participants) | 13
  PCS-12: Fistula With Low Intersphincteric Type- No | 43.93 (7.02)
  PCS-12: Fistula With Low Transsphincteric Type- Yes: number analyzed (Participants) | 3
  PCS-12: Fistula With Low Transsphincteric Type- Yes | 42.89 (7.61)
  PCS-12: Fistula With Low Transsphincteric Type- No: number analyzed (Participants) | 12
  PCS-12: Fistula With Low Transsphincteric Type- No | 45.98 (7.78)
  PCS-12: Fistula With Midline Position- Yes: number analyzed (Participants) | 11
  PCS-12: Fistula With Midline Position- Yes | 46.12 (8.04)
  PCS-12: Fistula With Midline Position- No: number analyzed (Participants) | 4
  PCS-12: Fistula With Midline Position- No | 43.26 (6.71)
  PCS-12: Fistula With Lateral Position- Yes: number analyzed (Participants) | 6
  PCS-12: Fistula With Lateral Position- Yes | 43.77 (6.43)
  PCS-12: Fistula With Lateral Position- No: number analyzed (Participants) | 9
  PCS-12: Fistula With Lateral Position- No | 46.42 (8.46)
  PCS-12: Fistula With Seton- Yes: number analyzed (Participants) | 8
  PCS-12: Fistula With Seton- Yes | 43.71 (4.71)
  PCS-12: Fistula With Seton- No: number analyzed (Participants) | 7
  PCS-12: Fistula With Seton- No | 47.25 (10.02)
  PCS-12: Harvey-Bradshaw Index (HBI) Category- Remission: number analyzed (Participants) | 12
  PCS-12: Harvey-Bradshaw Index (HBI) Category- Remission | 46.62 (7.93)
  PCS-12: HBI Category- Mild Activity: number analyzed (Participants) | 2
  PCS-12: HBI Category- Mild Activity | 38.85 (2.28)
  PCS-12: HBI Category- Moderate Activity: number analyzed (Participants) | 1
  PCS-12: HBI Category- Moderate Activity | 43.25 (NA) — Standard deviation (SD) was not estimable due to low number of participants with event.
  PCS-12: HBI Category- Severe Activity: number analyzed (Participants) | 0
  PCS-12: Treatment-naïve- Yes: number analyzed (Participants) | 1
  PCS-12: Treatment-naïve- Yes | 34.51 (NA) — Standard deviation (SD) was not estimable due to low number of participants with event.
  PCS-12: Treatment-naïve- No: number analyzed (Participants) | 14
  PCS-12: Treatment-naïve- No | 46.13 (7.23)
  PCS-12: Surgery-naïve- Yes: number analyzed (Participants) | 3
  PCS-12: Surgery-naïve- Yes | 37.93 (6.75)
  PCS-12: Surgery-naïve- No: number analyzed (Participants) | 12
  PCS-12: Surgery-naïve- No | 47.22 (6.79)
  PCS-12: Surgery - Fistulotomy- Yes: number analyzed (Participants) | 2
  PCS-12: Surgery - Fistulotomy- Yes | 45.08 (0.42)
  PCS-12: Surgery - Fistulotomy- No: number analyzed (Participants) | 13
  PCS-12: Surgery - Fistulotomy- No | 45.40 (8.19)
  PCS-12: Surgery - Advancement Flap- Yes: number analyzed (Participants) | 0
  PCS-12: Surgery - Advancement Flap- No | 45.36 (7.58)
  PCS-12: Surgery - Ligation of the Intersphincteric Fistula Tract (LIFT)- Yes: number analyzed (Participants) | 0
  PCS-12: Surgery - LIFT- No | 45.36 (7.58)
  PCS-12: Surgery - Fibrin Glue- Yes: number analyzed (Participants) | 0
  PCS-12: Surgery - Fibrin Glue- No | 45.36 (7.58)
  PCS-12: Surgery - Anal Fistula Plug- Yes: number analyzed (Participants) | 0
  PCS-12: Surgery - Anal Fistula Plug- No | 45.36 (7.58)
  PCS-12: Surgery - Defunctioning Stoma- Yes: number analyzed (Participants) | 0
  PCS-12: Surgery - Defunctioning Stoma- No | 45.36 (7.58)
  PCS-12: Surgery - Cutting Seton- Yes: number analyzed (Participants) | 0
  PCS-12: Surgery - Cutting Seton- No | 45.36 (7.58)
  PCS-12: Surgery - Loose Seton- Yes: number analyzed (Participants) | 9
  PCS-12: Surgery - Loose Seton- Yes | 46.56 (6.98)
  PCS-12: Surgery - Loose Seton- No: number analyzed (Participants) | 6
  PCS-12: Surgery - Loose Seton- No | 43.56 (8.76)
  PCS-12: Surgery - Other- Yes: number analyzed (Participants) | 4
  PCS-12: Surgery - Other- Yes | 47.28 (6.77)
  PCS-12: Surgery - Other- No: number analyzed (Participants) | 11
  PCS-12: Surgery - Other- No | 44.66 (8.05)
  PCS-12: Presence of Perianal Abscess- Yes: number analyzed (Participants) | 6
  PCS-12: Presence of Perianal Abscess- Yes | 47.57 (7.88)
  PCS-12: Presence of Perianal Abscess- No: number analyzed (Participants) | 9
  PCS-12: Presence of Perianal Abscess- No | 43.88 (7.47)
  PCS-12: Presence of Anorectal Stricture- Yes: number analyzed (Participants) | 0
  PCS-12: Presence of Anorectal Stricture- No | 45.36 (7.58)
Statistical Analysis 1: Comparison: CD Participants With CPF; PCS-12: Sex; Test type: Superiority; p = 0.1217, t-test for Independent Samples
Statistical Analysis 2: Comparison: CD Participants With CPF; PCS-12: Employment Status; Test type: Superiority; p = 0.8241, ANOVA; ANOVA=Analysis of variance
Statistical Analysis 3: Comparison: CD Participants With CPF; PCS-12: Smoking Status; Test type: Superiority; p = 0.3471, ANOVA
Statistical Analysis 4: Comparison: CD Participants With CPF; PCS-12: Age at Onset; Test type: Superiority; p = 0.9951, ANOVA
Statistical Analysis 5: Comparison: CD Participants With CPF; PCS-12: Disease Location; Test type: Superiority; p = 0.0631, ANOVA
Statistical Analysis 6: Comparison: CD Participants With CPF; PCS-12: Disease Behavior; Test type: Superiority; p = 0.7473, ANOVA
Statistical Analysis 7: Comparison: CD Participants With CPF; PCS-12: Presence of any Extraintestinal Manifestation of CD; Test type: Superiority; p = 0.4422, t-test for Independent Samples
Statistical Analysis 8: Comparison: CD Participants With CPF; PCS-12: Fistula With High Intersphincteric Type; Test type: Superiority; p = 0.1796, t-test for Independent Samples
Statistical Analysis 9: Comparison: CD Participants With CPF; PCS-12: Fistula With High Transsphincteric Type; Test type: Superiority; p = 0.3535, t-test for Independent Samples
Statistical Analysis 10: Comparison: CD Participants With CPF; PCS-12: Fistula With Suprasphincteric Type; Test type: Superiority; p = 0.1508, t-test for Independent Samples
Statistical Analysis 11: Comparison: CD Participants With CPF; PCS-12: Fistula with Extrasphincteric Type; Test type: Superiority; p = 0.2671, t-test for Independent Samples
Statistical Analysis 12: Comparison: CD Participants With CPF; PCS-12: Fistula With Low Intersphincteric Type; Test type: Superiority; p = 0.0594, t-test for Independent Samples
Statistical Analysis 13: Comparison: CD Participants With CPF; PCS-12: Fistula With Low Transsphincteric Type; Test type: Superiority; p = 0.5484, t-test for Independent Samples
Statistical Analysis 14: Comparison: CD Participants With CPF; PCS-12: Fistula With Midline Position; Test type: Superiority; p = 0.5387, t-test for Independent Samples
Statistical Analysis 15: Comparison: CD Participants With CPF; PCS-12: Fistula With Lateral Position; Test type: Superiority; p = 0.5270, t-test for Independent Samples
Statistical Analysis 16: Comparison: CD Participants With CPF; PCS-12: Fistula With Seton; Test type: Superiority; p = 0.3863, t-test for Independent Samples
Statistical Analysis 17: Comparison: CD Participants With CPF; PCS-12: HBI Categories (Remission, Mild and Moderate Activity); Test type: Superiority; p = 0.4206, ANOVA
Statistical Analysis 18: Comparison: CD Participants With CPF; PCS-12: Surgery-naïve; Test type: Superiority; p = 0.0538, t-test for Independent Samples
Statistical Analysis 19: Comparison: CD Participants With CPF; PCS-12: Surgery - Fistulotomy; Test type: Superiority; p = 0.9572, t-test for Independent Samples
Statistical Analysis 20: Comparison: CD Participants With CPF; PCS-12: Surgery - Loose Seton; Test type: Superiority; p = 0.4742, t-test for Independent Samples
Statistical Analysis 21: Comparison: CD Participants With CPF; PCS-12: Surgery - Other; Test type: Superiority; p = 0.5735, t-test for Independent Samples
Statistical Analysis 22: Comparison: CD Participants With CPF; PCS-12: Presence of Perianal Abscess; Test type: Superiority; p = 0.3760, t-test for Independent Samples

13. Secondary Outcome: Correlation Between General QoL MCS-12 and the Participants Socio-demographic, Anthropometric and Clinical Characteristics Assessed as MCS Score Stratified Based on Qualitative Variables
Description: The following qualitative variables were considered for the bivariate analysis: sex, smoking status, employment status, extraintestinal manifestations of Crohn's disease, Montreal classification for CD disease (age at onset, disease location, and disease behavior), fistula type and position, CD disease activity, treatment-naïve, surgery-naïve, type of surgery, and presence of seton, perianal abscess and anorectal stricture. MCS-12 scores were transformed to a 0 to 100, with higher scores indicating better quality of life.
Time Frame: At inclusion visit (Day 1)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CD Participants With CPF: Participants diagnosed with CD and Complex CPF in the Portuguese routine clinical practice were assessed. Retrospective data on healthcare resource utilization related with CPF management in the previous three years was obtained from the medical records.
Arm/Group | CD Participants With CPF
Number analyzed (Participants) | 15
score on a scale
  MCS-12: Sex- Male: number analyzed (Participants) | 7
  MCS-12: Sex- Male | 36.27 (5.60)
  MCS-12: Sex- Female: number analyzed (Participants) | 8
  MCS-12: Sex- Female | 39.51 (10.56)
  MCS-12: Employment Status- Employed: number analyzed (Participants) | 9
  MCS-12: Employment Status- Employed | 35.84 (9.17)
  MCS-12: Employment Status- Unemployed: number analyzed (Participants) | 3
  MCS-12: Employment Status- Unemployed | 41.22 (7.89)
  MCS-12: Employment Status- Retired: number analyzed (Participants) | 2
  MCS-12: Employment Status- Retired | 45.19 (3.63)
  MCS-12: Employment Status- Student: number analyzed (Participants) | 1
  MCS-12: Employment Status- Student | 33.45 (NA) — SD was not estimable due to low number of participants with event.
  MCS-12: Employment Status- Other: number analyzed (Participants) | 0
  MCS-12: Smoking Status- Never: number analyzed (Participants) | 8
  MCS-12: Smoking Status- Never | 38.54 (10.94)
  MCS-12: Smoking Status- Former: number analyzed (Participants) | 2
  MCS-12: Smoking Status- Former | 31.97 (2.62)
  MCS-12: Smoking Status- Current: number analyzed (Participants) | 5
  MCS-12: Smoking Status- Current | 39.55 (4.37)
  MCS-12: Age at Onset of CD Diagnosis- At or Below 16 Years: number analyzed (Participants) | 1
  MCS-12: Age at Onset of CD Diagnosis- At or Below 16 Years | 30.11 (NA) — SD was not estimable due to low number of participants with event.
  MCS-12: Age at Onset of CD Diagnosis- Between 17 and 40 Years: number analyzed (Participants) | 10
  MCS-12: Age at Onset of CD Diagnosis- Between 17 and 40 Years | 36.73 (8.55)
  MCS-12: Age at Onset of CD Diagnosis- Above 40 Years: number analyzed (Participants) | 4
  MCS-12: Age at Onset of CD Diagnosis- Above 40 Years | 43.16 (7.43)
  MCS-12: Disease Location 1- Terminal Ileum: number analyzed (Participants) | 4
  MCS-12: Disease Location 1- Terminal Ileum | 34.08 (13.03)
  MCS-12: Disease Location 1 + 4- Terminal Ileum + Upper Gastrointestinal: number analyzed (Participants) | 1
  MCS-12: Disease Location 1 + 4- Terminal Ileum + Upper Gastrointestinal | 33.45 (NA) — SD was not estimable due to low number of participants with event.
  MCS-12: Disease Location 2- Colon: number analyzed (Participants) | 3
  MCS-12: Disease Location 2- Colon | 46.18 (4.86)
  MCS-12: Disease Location 2 + 4- Colon + Upper Gastrointestinal: number analyzed (Participants) | 0
  MCS-12: Disease Location 3- Ileocolon: number analyzed (Participants) | 5
  MCS-12: Disease Location 3- Ileocolon | 39.58 (4.32)
  MCS-12: Disease Location 3 + 4- Ileocolon + Upper Gastrointestinal: number analyzed (Participants) | 2
  MCS-12: Disease Location 3 + 4- Ileocolon + Upper Gastrointestinal | 31.89 (2.52)
  MCS-12: Disease Location 4- Upper Gastrointestinal: number analyzed (Participants) | 0
  MCS-12: Disease Behavior- Nonstricturing, Nonpenetrating + Perianal: number analyzed (Participants) | 8
  MCS-12: Disease Behavior- Nonstricturing, Nonpenetrating + Perianal | 39.35 (7.19)
  MCS-12: Disease Behavior- Stricturing + Perianal: number analyzed (Participants) | 5
  MCS-12: Disease Behavior- Stricturing + Perianal | 34.05 (11.26)
  MCS-12: Disease Behavior- Penetrating + Perianal: number analyzed (Participants) | 2
  MCS-12: Disease Behavior- Penetrating + Perianal | 42.51 (2.35)
  MCS-12: Presence of any Extraintestinal Manifestation of CD- Yes: number analyzed (Participants) | 2
  MCS-12: Presence of any Extraintestinal Manifestation of CD- Yes | 38.80 (2.74)
  MCS-12: Presence of any Extraintestinal Manifestation of CD- No: number analyzed (Participants) | 13
  MCS-12: Presence of any Extraintestinal Manifestation of CD- No | 37.88 (9.12)
  MCS-12: Fistula With High Intersphincteric Type- Yes: number analyzed (Participants) | 3
  MCS-12: Fistula With High Intersphincteric Type- Yes | 37.64 (4.63)
  MCS-12: Fistula With High Intersphincteric Type- No: number analyzed (Participants) | 12
  MCS-12: Fistula With High Intersphincteric Type- No | 38.09 (9.36)
  MCS-12: Fistula With High Transsphincteric Type- Yes: number analyzed (Participants) | 3
  MCS-12: Fistula With High Transsphincteric Type- Yes | 37.23 (6.16)
  MCS-12: Fistula With High Transsphincteric Type- No: number analyzed (Participants) | 12
  MCS-12: Fistula With High Transsphincteric Type- No | 38.20 (9.19)
  MCS-12: Fistula With Suprasphincteric Type- Yes: number analyzed (Participants) | 2
  MCS-12: Fistula With Suprasphincteric Type- Yes | 45.46 (6.53)
  MCS-12: Fistula With Suprasphincteric Type- No: number analyzed (Participants) | 13
  MCS-12: Fistula With Suprasphincteric Type- No | 36.85 (8.35)
  MCS-12: Fistula With Extrasphincteric Type- Yes: number analyzed (Participants) | 2
  MCS-12: Fistula With Extrasphincteric Type- Yes | 40.71 (9.96)
  MCS-12: Fistula With Extrasphincteric Type- No: number analyzed (Participants) | 13
  MCS-12: Fistula With Extrasphincteric Type- No | 37.58 (8.62)
  MCS-12: Fistula With Superficial Type- Yes: number analyzed (Participants) | 0
  MCS-12: Fistula With Superficial Type- No | 38.00 (8.48)
  MCS-12: Fistula With Low Intersphincteric Type- Yes: number analyzed (Participants) | 2
  MCS-12: Fistula With Low Intersphincteric Type- Yes | 40.10 (14.47)
  MCS-12: Fistula With Low Intersphincteric Type- No: number analyzed (Participants) | 13
  MCS-12: Fistula With Low Intersphincteric Type- No | 37.68 (8.11)
  MCS-12: Fistula With Low Transsphincteric Type- Yes: number analyzed (Participants) | 3
  MCS-12: Fistula With Low Transsphincteric Type- Yes | 38.15 (5.38)
  MCS-12: Fistula With Low Transsphincteric Type- No: number analyzed (Participants) | 12
  MCS-12: Fistula With Low Transsphincteric Type- No | 37.96 (9.29)
  MCS-12: Fistula With Midline Position- Yes: number analyzed (Participants) | 11
  MCS-12: Fistula With Midline Position- Yes | 39.59 (7.05)
  MCS-12: Fistula With Midline Position- No: number analyzed (Participants) | 4
  MCS-12: Fistula With Midline Position- No | 33.63 (11.63)
  MCS-12: Fistula With Lateral Position- Yes: number analyzed (Participants) | 6
  MCS-12: Fistula With Lateral Position- Yes | 36.33 (9.95)
  MCS-12: Fistula With Lateral Position- No: number analyzed (Participants) | 9
  MCS-12: Fistula With Lateral Position- No | 39.12 (7.78)
  MCS-12: Fistula With Seton- Yes: number analyzed (Participants) | 8
  MCS-12: Fistula With Seton- Yes | 36.36 (9.36)
  MCS-12: Fistula With Seton- No: number analyzed (Participants) | 7
  MCS-12: Fistula With Seton- No | 39.87 (7.63)
  MCS-12: HBI Category- Remission: number analyzed (Participants) | 12
  MCS-12: HBI Category- Remission | 37.15 (8.66)
  MCS-12: HBI Category- Mild Activity: number analyzed (Participants) | 2
  MCS-12: HBI Category- Mild Activity | 45.40 (6.60)
  MCS-12: HBI Category- Moderate Activity: number analyzed (Participants) | 1
  MCS-12: HBI Category- Moderate Activity | 33.45 (NA) — SD was not estimable due to low number of participants with event.
  MCS-12: HBI Category- Severe Activity: number analyzed (Participants) | 0
  MCS-12: Treatment-naïve- Yes: number analyzed (Participants) | 1
  MCS-12: Treatment-naïve- Yes | 36.47 (NA) — SD was not estimable due to low number of participants with event.
  MCS-12: Treatment-naïve- No: number analyzed (Participants) | 14
  MCS-12: Treatment-naïve- No | 38.11 (8.79)
  MCS-12: Surgery-naïve- Yes: number analyzed (Participants) | 3
  MCS-12: Surgery-naïve- Yes | 39.30 (7.45)
  MCS-12: Surgery-naïve- No: number analyzed (Participants) | 12
  MCS-12: Surgery-naïve- No | 37.68 (9.00)
  MCS-12: Surgery - Fistulotomy- Yes: number analyzed (Participants) | 2
  MCS-12: Surgery - Fistulotomy- Yes | 31.97 (2.62)
  MCS-12: Surgery - Fistulotomy- No: number analyzed (Participants) | 13
  MCS-12: Surgery - Fistulotomy- No | 38.93 (8.74)
  MCS-12: Surgery - Advancement Flap- Yes: number analyzed (Participants) | 0
  MCS-12: Surgery - Advancement Flap- No | 38.00 (8.48)
  MCS-12: Surgery - Ligation of the Intersphincteric Fistula Tract (LIFT) - Yes: number analyzed (Participants) | 0
  MCS-12: Surgery - LIFT- No | 38.00 (8.48)
  MCS-12: Surgery - Fibrin Glue- Yes: number analyzed (Participants) | 0
  MCS-12: Surgery - Fibrin Glue- No | 38.00 (8.48)
  MCS-12: Surgery - Anal Fistula Plug- Yes: number analyzed (Participants) | 0
  MCS-12: Surgery - Anal Fistula Plug- No | 38.00 (8.48)
  MCS-12: Surgery - Defunctioning Stoma- Yes: number analyzed (Participants) | 0
  MCS-12: Surgery - Defunctioning Stoma- No | 38.00 (8.48)
  MCS-12: Surgery - Cutting Seton-Yes: number analyzed (Participants) | 0
  MCS-12: Surgery - Cutting Seton- No | 38.00 (8.48)
  MCS-12: Surgery - Loose Seton- Yes: number analyzed (Participants) | 9
  MCS-12: Surgery - Loose Seton- Yes | 39.81 (9.46)
  MCS-12: Surgery - Loose Seton- No: number analyzed (Participants) | 6
  MCS-12: Surgery - Loose Seton- No | 35.28 (6.60)
  MCS-12: Surgery - Other- Yes: number analyzed (Participants) | 4
  MCS-12: Surgery - Other- Yes | 46.80 (3.98)
  MCS-12: Surgery - Other- No: number analyzed (Participants) | 11
  MCS-12: Surgery - Other- No | 34.80 (7.34)
  MCS-12: Presence of Perianal Abscess- Yes: number analyzed (Participants) | 6
  MCS-12: Presence of Perianal Abscess- Yes | 35.59 (10.91)
  MCS-12: Presence of Perianal Abscess- No: number analyzed (Participants) | 9
  MCS-12: Presence of Perianal Abscess- No | 39.61 (6.65)
  MCS-12: Presence of Anorectal Stricture- Yes: number analyzed (Participants) | 0
  MCS-12: Presence of Anorectal Stricture- No | 38.00 (8.48)
Statistical Analysis 1: Comparison: CD Participants With CPF; MCS-12: Sex; Test type: Superiority; p = 0.4814, t-test for Independent Samples
Statistical Analysis 2: Comparison: CD Participants With CPF; MCS-12: Employment Status; Test type: Superiority; p = 0.3136, Kruskal-Wallis
Statistical Analysis 3: Comparison: CD Participants With CPF; MCS-12: Smoking Status; Test type: Superiority; p = 0.5808, ANOVA
Statistical Analysis 4: Comparison: CD Participants With CPF; MCS-12: Age at Onset; Test type: Superiority; p = 0.2965, ANOVA
Statistical Analysis 5: Comparison: CD Participants With CPF; MCS-12: Disease Location; Test type: Superiority; p = 0.2874, ANOVA
Statistical Analysis 6: Comparison: CD Participants With CPF; MCS-12: Disease Behavior; Test type: Superiority; p = 0.4269, ANOVA
Statistical Analysis 7: Comparison: CD Participants With CPF; MCS-12: Presence of any Extraintestinal Manifestation of CD; Test type: Superiority; p = 0.8931, t-test for Independent Samples
Statistical Analysis 8: Comparison: CD Participants With CPF; MCS-12: Fistula With High Intersphincteric Type; Test type: Superiority; p = 0.9384, t-test for Independent Samples
Statistical Analysis 9: Comparison: CD Participants With CPF; MCS-12: Fistula With High Transsphincteric Type; Test type: Superiority; p = 0.8286, Mann-Whitney
Statistical Analysis 10: Comparison: CD Participants With CPF; MCS-12: Fistula With Suprasphincteric Type; Test type: Superiority; p = 0.1919, t-test for Independent Samples
Statistical Analysis 11: Comparison: CD Participants With CPF; MCS-12: Fistula with Extrasphincteric Type; Test type: Superiority; p = 0.6452, t-test for Independent Samples
Statistical Analysis 12: Comparison: CD Participants With CPF; MCS-12: Fistula With Low Intersphincteric Type; Test type: Superiority; p = 0.7218, t-test for Independent Samples
Statistical Analysis 13: Comparison: CD Participants With CPF; MCS-12: Fistula With Low Transsphincteric Type; Test type: Superiority; p = 0.9738, t-test for Independent Samples
Statistical Analysis 14: Comparison: CD Participants With CPF; MCS-12: Fistula With Midline Position; Test type: Superiority; p = 0.2419, t-test for Independent Samples
Statistical Analysis 15: Comparison: CD Participants With CPF; MCS-12: Fistula With Lateral Position; Test type: Superiority; p = 0.5524, t-test for Independent Samples
Statistical Analysis 16: Comparison: CD Participants With CPF; MCS-12: Fistula With Seton; Test type: Superiority; p = 0.4443, t-test for Independent Samples
Statistical Analysis 17: Comparison: CD Participants With CPF; MCS-12: HBI Categories (Remission, Mild and Moderate Activity); Test type: Superiority; p = 0.4106, ANOVA
Statistical Analysis 18: Comparison: CD Participants With CPF; MCS-12: Surgery-naïve; Test type: Superiority; p = 0.7795, t-test for Independent Samples
Statistical Analysis 19: Comparison: CD Participants With CPF; MCS-12: Surgery - Fistulotomy; Test type: Superiority; p = 0.2964, t-test for Independent Samples
Statistical Analysis 20: Comparison: CD Participants With CPF; MCS-12: Surgery - Loose Seton; Test type: Superiority; p = 0.3287, t-test for Independent Samples
Statistical Analysis 21: Comparison: CD Participants With CPF; MCS-12: Surgery - Other; Test type: Superiority; p = 0.0091, t-test for Independent Samples
Statistical Analysis 22: Comparison: CD Participants With CPF; MCS-12: Presence of Perianal Abscess; Test type: Superiority; p = 0.3889, t-test for Independent Samples

14. Secondary Outcome: Correlation Between General QoL PCS-12 and the Participants Socio-demographic, Anthropometric and Clinical Characteristics Assessed as Correlation Coefficient Stratified Based on Quantitative Variables
Description: The following quantitative variables were considered for bivariate analysis: age, BMI, time between CD diagnosis date and date of study visit, total number of CPFs per participant, time between first CPF diagnosis date and date of study visit, Perianal Disease Activity Index (PDAI) score, number of internal and external fistula openings, time since seton placement, SIBDQ score, SQoL-M score (for male participants) and SQoL-F score (for female participants), and Wexner score. Data was collected and reported as number for all the quantitative variables as the associations (correlation coefficient) between general QoL and the quantitative variables was calculated using Spearman Correlation Coefficients.
Time Frame: At inclusion visit (Day 1)
Population: as for outcome 7
Measure: Number; unit: correlation coefficient
Arm/Group | CD Participants With CPF
Number analyzed (Participants) | 15
correlation coefficient
  PCS- 12: Age | -0.072
  PCS- 12: BMI | 0.210
  PCS- 12: Time Between CD Diagnosis Date and Date of Study Visit | -0.014
  PCS- 12: Total Number of CPFs per Participant | -0.270
  PCS- 12: Time Since Seton Placement: number analyzed (Participants) | 9
  PCS- 12: Time Since Seton Placement | -0.185
  PCS- 12: Time Between First CPF Diagnosis Date and Date of Study Visit | 0.071
  PCS- 12: PDAI Score | -0.707
  PCS - 12: Number of Internal Fistula Openings per Participant | -0.450
  PCS- 12: Number of External Fistula Openings per Participant | -0.442
  PCS- 12: SIBDQ Score | 0.525
  PCS- 12: SQoL-M Score: number analyzed (Participants) | 7
  PCS- 12: SQoL-M Score | 0.690
  PCS- 12: SQoL-F Score: number analyzed (Participants) | 5
  PCS- 12: SQoL-F Score | 0.046
  PCS- 12: Wexner Score: number analyzed (Participants) | 14
  PCS- 12: Wexner Score | -0.259
Statistical Analysis 1: Comparison: CD Participants With CPF; PCS- 12: Age; Test type: Superiority; p = 0.8001, Pearson Correlation Coefficient
Statistical Analysis 2: Comparison: CD Participants With CPF; PCS- 12: BMI; Test type: Superiority; p = 0.4532, Pearson Correlation Coefficient
Statistical Analysis 3: Comparison: CD Participants With CPF; PCS- 12: Time Between CD Diagnosis Date and Date of Study Visit; Test type: Superiority; p = 0.9597, Spearman Correlation Coefficient
Statistical Analysis 4: Comparison: CD Participants With CPF; PCS- 12: Total Number of CPFs per Participant; Test type: Superiority; p = 0.3304, Spearman Correlation Coefficient
Statistical Analysis 5: Comparison: CD Participants With CPF; PCS- 12: Time Since Seton Replacement; Test type: Superiority; p = 0.6333, Pearson Correlation Coefficient
Statistical Analysis 6: Comparison: CD Participants With CPF; PCS- 12: Time Between First CPF Diagnosis Date and Date of Study Visit; Test type: Superiority; p = 0.8003, Spearman Correlation Coefficient
Statistical Analysis 7: Comparison: CD Participants With CPF; PCS- 12: PDAI Score; Test type: Superiority; p = 0.0032, Pearson Correlation Coefficient
Statistical Analysis 8: Comparison: CD Participants With CPF; PCS- 12: Number of Internal Fistula Openings per Participant; Test type: Superiority; p = 0.0923, Spearman Correlation Coefficient
Statistical Analysis 9: Comparison: CD Participants With CPF; PCS- 12: Number of External Fistula Openings per Participant; Test type: Superiority; p = 0.0994, Spearman Correlation Coefficient
Statistical Analysis 10: Comparison: CD Participants With CPF; PCS- 12: SIBDQ Score; Test type: Superiority; p = 0.0444, Pearson Correlation Coefficient
Statistical Analysis 11: Comparison: CD Participants With CPF; PCS- 12: SQoL-M Score; Test type: Superiority; p = 0.0860, Pearson Correlation Coefficient
Statistical Analysis 12: Comparison: CD Participants With CPF; PCS- 12: SQoL-F Score; Test type: Superiority; p = 0.9415, Pearson Correlation Coefficient
Statistical Analysis 13: Comparison: CD Participants With CPF; PCS- 12: Wexner Score; Test type: Superiority; p = 0.3709, Pearson Correlation Coefficient

15. Secondary Outcome: Correlation Between General QoL MCS-12 and the Participants Socio-demographic, Anthropometric and Clinical Characteristics Assessed as Correlation Coefficient Stratified Based on Quantitative Variables
Description: The following quantitative variables were considered for bivariate analysis: age, BMI, time between CD diagnosis date and date of study visit, total number of CPFs per participant, time between first CPF diagnosis date and date of study visit, PDAI score, number of internal and external fistula openings, time since seton placement, SIBDQ score, SQoL-M score (for male participants) and SQoL-F score (for female participants), and Wexner score. Data was collected and reported as number for all the quantitative variables as the associations (correlation coefficient) between general QoL and the quantitative variables was calculated using Spearman Correlation Coefficients.
Time Frame: At inclusion visit (Day 1)
Population: as for outcome 7
Measure: Number; unit: correlation coefficient
Arm/Group | CD Participants With CPF
Number analyzed (Participants) | 15
correlation coefficient
  MCS- 12: Age | 0.484
  MCS- 12: BMI | 0.022
  MCS- 12: Time Between CD Diagnosis Date and Date of Study Visit | -0.132
  MCS- 12: Total Number of CPFs per Participant | 0.077
  MCS- 12: Time Since Seton Placement: number analyzed (Participants) | 9
  MCS- 12: Time Since Seton Placement | -0.323
  MCS- 12: Time Between First CPF Diagnosis Date and Date of Study Visit | -0.018
  MCS- 12: PDAI Score | 0.067
  MCS- 12: Number of Internal Fistula Openings per Participant | -0.207
  MCS- 12: Number of External Fistula Openings per Participant | -0.048
  MCS- 12: SIBDQ Score | 0.404
  MCS- 12: SQoL-M Score: number analyzed (Participants) | 7
  MCS- 12: SQoL-M Score | 0.266
  MCS- 12: SQoL-F Score: number analyzed (Participants) | 5
  MCS- 12: SQoL-F Score | 0.039
  MCS- 12: Wexner Score: number analyzed (Participants) | 14
  MCS- 12: Wexner Score | -0.182
Statistical Analysis 1: Comparison: CD Participants With CPF; MCS- 12: Age; Test type: Superiority; p = 0.0674, Pearson Correlation Coefficient
Statistical Analysis 2: Comparison: CD Participants With CPF; MCS- 12: BMI; Test type: Superiority; p = 0.9392, Pearson Correlation Coefficient
Statistical Analysis 3: Comparison: CD Participants With CPF; MCS- 12: Time Between CD Diagnosis Date and Date of Study Visit; Test type: Superiority; p = 0.6387, Spearman Correlation Coefficient
Statistical Analysis 4: Comparison: CD Participants With CPF; MCS- 12: Total Number of CPFs per Participant; Test type: Superiority; p = 0.7846, Spearman Correlation Coefficient
Statistical Analysis 5: Comparison: CD Participants With CPF; MCS- 12: Time Since Seton Placement; Test type: Superiority; p = 0.3972, Pearson Correlation Coefficient
Statistical Analysis 6: Comparison: CD Participants With CPF; MCS- 12: Time Between First CPF Diagnosis Date and Date of Study Visit; Test type: Superiority; p = 0.9496, Spearman Correlation Coefficient
Statistical Analysis 7: Comparison: CD Participants With CPF; MCS- 12: PDAI Score; Test type: Superiority; p = 0.8130, Pearson Correlation Coefficient
Statistical Analysis 8: Comparison: CD Participants With CPF; MCS- 12: Number of Internal Fistula Openings per Participant; Test type: Superiority; p = 0.4588, Spearman Correlation Coefficient
Statistical Analysis 9: Comparison: CD Participants With CPF; MCS- 12: Number of External Fistula Openings per Participant; Test type: Superiority; p = 0.8663, Spearman Correlation Coefficient
Statistical Analysis 10: Comparison: CD Participants With CPF; MCS- 12: SIBDQ Score; Test type: Superiority; p = 0.1349, Pearson Correlation Coefficient
Statistical Analysis 11: Comparison: CD Participants With CPF; MCS- 12: SQoL-M Score; Test type: Superiority; p = 0.5647, Pearson Correlation Coefficient
Statistical Analysis 12: Comparison: CD Participants With CPF; MCS- 12: SQoL-F Score; Test type: Superiority; p = 0.9509, Pearson Correlation Coefficient
Statistical Analysis 13: Comparison: CD Participants With CPF; MCS- 12: Wexner Score; Test type: Superiority; p = 0.5328, Pearson Correlation Coefficient

ADVERSE EVENTS:
Time Frame: Up to 10 months 18 days
Arm/Group | CD Participants With CPF
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT04876690/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/90/NCT04876690/SAP_001.pdf